CLINICAL TRIAL: NCT07059858
Title: Evaluation of Bladder and Bowel Functions, Participation and Quality of Life in Children With Intellectual Disabilities
Brief Title: Bladder and Bowel Functions, Participation and Quality of Life in Children With Intellectual Disabilities
Status: Recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Other Study IDs: AIBU-FTR-ST-06
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Intellectual Disability; Healthy Subjects
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intellectual Disability Group: Individuals between the ages of 5-12 years with a diagnosis of intellectual disability
- Typical Developing Group: Typically developing individuals between the ages of 5-12

SUMMARY:
Many neurodevelopmental, psychiatric, and medical disorders are commonly associated with intellectual disability. The presence of neurodevelopmental and psychiatric (NDP) comorbidities has been reported to negatively impact the clinical outcomes of bowel or bladder dysfunction.

Pediatric bladder and bowel dysfunction (BBD) is a common but underdiagnosed condition characterized by a spectrum of lower urinary tract symptoms and is often associated with constipation. Lower urinary tract symptoms include dysuria, urinary urgency, daytime incontinence, and enuresis, while bowel symptoms include constipation and encopresis. Most BBD cases are functional and not neurogenic in origin.

In children with special needs, all types of urinary incontinence are reported to occur more frequently compared to children without developmental or behavioral disabilities. Intellectual disability (IQ <70) is also identified as a significant risk factor for urinary incontinence, with prevalence increasing as IQ decreases. In these children, lower urinary tract symptoms such as overactive bladder, dysfunctional voiding, and low fluid intake are also observed. Furthermore, according to support plans and medical records, 94% of individuals with intellectual and multiple disabilities experience constipation. Interestingly, lower levels of intellectual disability (profound and severe ID) have been associated with a lower prevalence of constipation.

Although there are studies in the literature examining bladder and bowel functions separately in specific diagnostic groups with intellectual disability, the number of studies that assess bladder and bowel functions together in children with any form of intellectual disability is limited. Moreover, to our knowledge, there is no study in the literature that evaluates bladder and bowel functions along with child participation and parental quality of life in children with intellectual disability.

Based on this gap in the literature, the aim of our study is to examine bladder and bowel functions, participation, and quality of life in children with intellectual disability

DETAILED DESCRIPTION:
This cross-sectional study will include children aged 5-12 years with intellectual disabilities who are attending Special Education and Rehabilitation Centers, as well as typically developing children. Necessary approvals will be obtained from the Non-Interventional Clinical Research Ethics Committee of Bolu Abant Izzet Baysal University.

Participants will be selected according to predefined inclusion criteria. Informed consent will be obtained from both the children included in the study and their parents. Sociodemographic data such as parents' age, height, weight, marital status, and education level will be recorded. Similarly, data on the children, including age, height, weight, and gender, will be collected.

Bladder and bowel functions of the children included in the study will be assessed using the Childhood Bladder and Bowel Dysfunction Questionnaire (CBBDQ), the Dysfunctional Voiding and Incontinence Scoring System (DVISS), and the Lower Urinary Tract Symptom Score (LUTSS). Child participation will be evaluated using the Child and Adolescent Scale of Participation (CASP). Parental quality of life will be assessed using the Nottingham Health Profile (NHP), and children's quality of life will be evaluated using the Pediatric Quality of Life Inventory - Gastrointestinal Symptoms Module (PedsQL GI Module)

ELIGIBILITY:
Inclusion Criteria:

For Children with Intellectual Disabilities:

* Aged between 5 and 12 years
* Diagnosed with mild, moderate, or severe intellectual disability as documented by the ÇÖZGER (Child Special Needs Report)
* Both the parent and the child agree to participate in the study

For Typically Developing Children

* Aged between 5 and 12 years
* Both the parent and the child agree to participate in the study

Exclusion Criteria:

For Children with Intellectual Disabilities:

* Having a diagnosis of physical disability
* Presence of a neurological anomaly affecting bladder and bowel functions
* Parent does not consent to participate in the study
* Having undergone trauma or surgery affecting bladder and bowel functions within the last 6 months
* Diagnosis of a genetic disorder
* Use of medications that may affect bladder and bowel functions

For Typically Developing Children

* Presence of a neurological anomaly affecting bladder and bowel functions
* Lack of parental consent to participate in the study
* Having experienced trauma or undergone surgery affecting bladder and bowel functions within the past 6 months
* Use of medications that may influence bladder and bowel functions

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Children diagnosed with intellectual disability and typically developing peers who agreed to participate in the study and met the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Childhood Bladder and Bowel Dysfunction Questionnaire (CBBDQ | baseline
  The CBBDQ is a parent-reported instrument used to assess and quantitatively measure symptoms of bladder and bowel dysfunction in children. It is designed for children aged 5 to 12 years and consists of 18 items, including 10 items related to bladder symptoms and 8 items related to bowel symptoms. Each item is rated on a five-point Likert scale ranging from 0 (never) to 4 (almost every day or every day). Higher CBBDQ scores indicate the presence of more severe or frequent symptoms.
Bladder and Bowel Dysfunction Scale (BBDS) | baseline
  The BBDS is a 14-item questionnaire designed to assess pediatric bladder and bowel dysfunction. Each item is rated using a five-point Likert scale. The total score ranges from 0 to 52, with higher scores indicating greater symptom severity. The scale includes 14 questions, of which the first 13 specifically address symptoms related to bladder and bowel dysfunction. The final question evaluates the level of difficulty experienced while completing the questionnaire and is not included in the total score.
Voiding Dysfunction Symptom Score (VDSS) | baseline
  The Voiding Dysfunction Symptom Score (VDSS) was developed by Akbal et al. in 2005 and consists of 14 items. Thirteen of the items assess symptoms related to daytime urinary incontinence, nighttime urinary incontinence (enuresis), urinary frequency during the day, the presence of constipation, and various lower urinary tract symptoms. The 14th item evaluates the impact of these symptoms on quality of life.
  The total score ranges from 0 to 35 points, with higher scores indicating increased severity of voiding dysfunction symptoms. The overall score is considered to be 35+3, with the additional 3 points referring to the quality-of-life impact assessment.
Child and Adolescent Scale of Participation (CASP) | baseline
  The Child and Adolescent Scale of Participation (CASP) is a caregiver-reported measure used to assess the extent to which school-aged children (aged 5 years and older) participate in home, school, and community activities compared to their same-age peers. The scale consists of 20 items grouped into four subdomains: Home Participation (6 items), Community Participation (4 items), School Participation (5 items), and Home and Community Living Activities (5 items).
  Each of the 20 items is rated on a four-point scale: "Age Expected (Full participation)," "Somewhat Limited," "Very Limited," and "Unable to Participate." If the item reflects an activity that is not age-appropriate for the child (e.g., employment), the response "Not Applicable" is selected. Higher scores indicate greater levels of participation.
  In addition, the CASP includes five open-ended questions that explore effective strategies and supports, as well as barriers that may influence the child's participation.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory - Gastrointestinal Symptoms Module (PedsQL GI Module) | baseline
  The PedsQL GI Module is designed for different age groups (2-4 years, 5-7 years, 8-12 years, and 13-18 years). It includes 74 items for both child self-report and parent proxy-report versions. The module consists of 10 separate Likert-type subscales that assess various gastrointestinal symptoms. Higher scores on the PedsQL GI Module indicate better health-related quality of life, while lower scores reflect a greater negative impact of gastrointestinal symptoms on quality of life.
Nottingham Health Profile (NHP) | baseline
  The Nottingham Health Profile (NHP) is used to assess health-related quality of life. It is a general quality of life questionnaire that measures an individual's perceived health problems and the extent to which these problems affect normal daily activities. The questionnaire consists of 38 items and evaluates six dimensions of health status. The items are answered with a "yes" or "no" response. Each section is scored on a scale from 0 to 100, where a score of 0 indicates the best possible health status and a score of 100 indicates the worst. Within the scope of this study, both the subscale scores and the total NHP score will be evaluated. The total NHP score will be calculated as the sum of the subscale scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sezen Tezcan, PhD, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University Faculty of Health Science, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No